CLINICAL TRIAL: NCT06132490
Title: Comparison of the Perioperative Effects of Intra-abdominal Pressure Created With Standard and Valveless Insufflators in Robotic Surgery
Brief Title: Intra-abdominal Pressure and Insufflator Effects in Robotic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2022.094.IRB1.040
Record Dates: First submitted 2023-03-20; First posted 2023-11-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-09

CONDITIONS: Post Operative Pain; Hemodynamic Instability; Hypercapnia; Complication,Postoperative; Intraoperative Complications
Keywords: robotic surgery; intra-abdominal pressure; insufflator; postoperative pain; postoperative complications; intraoperative complications
MeSH Terms: conditions — Pain, Postoperative; Hypercapnia; Postoperative Complications; Intraoperative Complications

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patient and the pain nurses will be blind to the intervention due to the study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Valveless 12 (Experimental): Patients scheduled for genitourinary or colorectal robotic surgery, valveless insufflators will be used with 12 mmHg intra-abdominal pressure.
  Interventions: Device: Valveless Insufflator with 12 mmHg intra-abdominal pressure
- Valveless 8 (Experimental): Patients scheduled for genitourinary or colorectal robotic surgery, valveless insufflators will be used with 8 mmHg intra-abdominal pressure.
  Interventions: Device: Valveless Insufflator with 8 mmHg intra-abdominal pressure

INTERVENTIONS:
Device: Valveless Insufflator with 12 mmHg intra-abdominal pressure — In this group valveless insufflators, which are relatively new in clinical practice, will be used under low intra-abdominal pressure throughout the surgery.
  Arms: Valveless 12
Device: Valveless Insufflator with 8 mmHg intra-abdominal pressure — In this group valveless insufflators, which are relatively new in clinical practice, will be used under ultra-low intra-abdominal pressure throughout the surgery.
  Arms: Valveless 8

SUMMARY:
The main aim of this study is to compare the perioperative effects of different intra-abdominal pressures and different insufflators in patients undergoing robotic surgery at a 30-45 degree trendelenburg position.

DETAILED DESCRIPTION:
Adult patients scheduled for robotic genitourinary or colorectal surgery are going to be enrolled in this study. Patients will be randomized in three groups. In group I, conventional insufflators will be used with 12 mmHg intra-abdominal pressure; in group II, valveless insufflators will be used with 12 mmHg intra-abdominal pressure and in group III, valveless insufflators will be used with 8 mmHg intra-abdominal pressure. Intraoperative data regarding airway pressures, lung compliance, hemodynamic parameters, arterial blood gas analysis, times of pressure loss and camera cleaning will be gathered. Each patient will receive a standardized anesthesia and analgesia procedure with a intravenous morphine patient controlled analgesia (PCA). Postoperative pain will be monitored at 1st, 3rd, 6th, 12th and 24th postoperative hours and morphine consumption rates will be recorded. Patient length of stay, time to first flatus, urine output, postoperative complications(graded by Clavien Dindo classification), preoperative and postoperative hemoglobin and creatinine levels will be filed.

ELIGIBILITY:
Inclusion Criteria:

* Elective robotic surgery with intraabdominal insufflation and trendelenburg position (prostatectomy, hemicolectomy etc.)
* ASA (American Society of Anesthesiologists) Physical Status I-II-III

Exclusion Criteria:

* Patients without consent
* Emergency surgery
* Bleeding diathesis
* Pregnancy or lactation
* Prior history of major abdominal/pelvic surgery
* Chronic kidney disease
* Chronic opioid consumption for chronic pain
* Inability to communicate with the patient due to language barriers or mental status

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Number of manipulations done by the attending anesthesiologists | Intraoperative
  After the induction of general anesthesia, orotracheal intubation and arterial catheterization; a standard ventilation and anesthesia maintenance strategy will be applied. Every manipulation performed to keep the parameters monitored by the anesthesiologists within physiological limits will be recorded: ventilation frequency setting, remifentail infusion titration, administration of vasoactive agents, etc.

SECONDARY OUTCOMES:
Arterial blood gas lactate levels | Intraoperative
  Arterial blood gas will be sampled at standardized times during the operation and lactate levels will be compared among the groups
Peak airway pressures | Intraoperative
  Peak airway pressures (cmH2O) will be compared among the groups
Mean airway pressures | Intraoperative
  Mean airway pressures (cmH2O) will be compared among the groups
Lung compliance | Intraoperative
  Lung compliance (mL/cmH2O) will be compared among the groups
End tidal carbon dioxide levels | Intraoperative
  End tidal carbon dioxide levels (mmHg) will be compared among the groups
Minute ventilation | Intraoperative
  Minute ventilation (L/minute) will be compared among the groups
Systolic blood pressure | Intraoperative
  Systolic arterial pressures (mmHg) will be compared among the groups.
Diastolic blood pressure | Intraoperative
  Diastolic arterial pressures (mmHg) will be compared among the groups.
Mean blood pressure | Intraoperative
  Mean arterial pressures (mmHg) will be compared among the groups.
Heart rate | Intraoperative
  Heart rate (beat per minute) will be compared among the groups
Acute Postoperative Pain | Postoperative 24 hours
  Acute postoperative pain reported with numeric rating scale (0-10) will be recorded at postoperative 1st, 3rd, 6th, 12th and 24th hours with 0 meaning no pain and 10 meaning worst imaginable pain.
Postoperative morphine consumption | Postoperative 24 hours
  Intravenous morphine consumption (mg) will be recorded at postoperative 1st, 3rd, 6th, 12th and 24th hours
Anesthesia time and operative time | Intraoperative
  Anesthesia and operative times wil be recorded as minutes
Intraoperative bleeding | Intraoperative
  Total bleeding level estimated by the surgical nurse will be recorded as milliliters at the end of the surgery
Urine output | Intraoperative and daily untill discharge
  Kidney function will be monitored by using intraoperative and daily postoperative urine output (mL)
Creatinine levels | Preoperative and postoperative (up to one month)
  Kidney function will be monitored by using daily creatinine levels (mg/dL)
Hemoglobin levels | Intraoperative and daily untill discharge
  Intraoperative and daily postoperative hemoglobin levels will be recorded
Need for blood product transfusion | Intraoperative and daily untill discharge
  Blood product transfusions will be recorded
Number of participants with pulmonary complications | Postoperative, up to one month
  Pulmonary complications like atelectasis, pulmonary oedema, pleural effusion, pneumothorax, pneumonia, ventilatory failure will be recorded for each patient. And number of patients with pulmonary complications will be compared among the groups.
Flatus time | Postoperative one week
  Postoperative time to first flatus will be recorded
Time to oral intake | Postoperative 3 days
  Postoperative time to oral intake will be recorded
Number of participants with subcutaneous emphysema | Postoperative, up to one month
  Subcutaneous emphysema diagnosed with chest radiograph will be recorded
Length of hospital stay | Postoperative, up to one month
  Length of hospital stay will be recorded as hours
The Clavien-Dindo classification of surgical complications | Postoperative, up to one month
  Any postoperative complication will be graded by the Clavien-Dindo classification between I to V with I meaning any deviation from the postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions and V meaning death of a patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Koç University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data collected for the study, including de-identified individual participant data will be made available to other within 6 months after the publication of this trial, as will additional related documents (study protocol, statistical analysis plan and informed consent form), for academic purposes (e.g , meta-analyses) upon request to the corresponding author, and with a signed data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after the publication
Access Criteria: Academic purposes

REFERENCES:
- [Background] Feng TS, Heulitt G, Islam A, Porter JR. Comparison of valve-less and standard insufflation on pneumoperitoneum-related complications in robotic partial nephrectomy: a prospective randomized trial. J Robot Surg. 2021 Jun;15(3):381-388. doi: 10.1007/s11701-020-01117-z. Epub 2020 Jul 6. PMID 32632561
- [Background] Horstmann M, Horton K, Kurz M, Padevit C, John H. Prospective comparison between the AirSeal(R) System valve-less Trocar and a standard Versaport Plus V2 Trocar in robotic-assisted radical prostatectomy. J Endourol. 2013 May;27(5):579-82. doi: 10.1089/end.2012.0632. Epub 2013 Feb 5. PMID 23186377
- [Background] Paull JO, Parsacandola SA, Graham A, Hota S, Pudalov N, Obias V. The impact of the AirSeal(R) valve-less trocar system in robotic colorectal surgery: a single-surgeon retrospective review. J Robot Surg. 2021 Feb;15(1):87-92. doi: 10.1007/s11701-020-01071-w. Epub 2020 Apr 24. PMID 32333365
- [Background] La Falce S, Novara G, Gandaglia G, Umari P, De Naeyer G, D'Hondt F, Beresian J, Carette R, Penicka M, Mo Y, Vandenbroucke G, Mottrie A. Low Pressure Robot-assisted Radical Prostatectomy With the AirSeal System at OLV Hospital: Results From a Prospective Study. Clin Genitourin Cancer. 2017 Dec;15(6):e1029-e1037. doi: 10.1016/j.clgc.2017.05.027. Epub 2017 Jun 2. PMID 28669704